CLINICAL TRIAL: NCT05719831
Title: Optimization of Vonoprazan--amoxicillin Dual Therapy for Eradicating Helicobacter pyloriinfection-a Multicenter, Prospective, Randomized, Parallel-controlled Study
Brief Title: Optimization of Vonoprazan--amoxicillin Dual Therapy for Eradicating Helicobacter Pyloriinfection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Peng, Attending physician, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Eradication Rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- H-VA-dual-10 (Experimental): 10 days(vonoprazan fumarate tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 750mg/ time, 4 times/day, oral)
  Interventions: Drug: vonoprazan fumarate + high dose amoxicillin（H-10d）
- L-VA-dual-10 (Experimental): 10 days(vonoprazan fumarate tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 1000mg/ time, 2 times/day, oral)
  Interventions: Drug: vonoprazan fumarate + low dose amoxicillin（L-10d)
- H-VA-dual-14 (Active Comparator): 14 days(vonoprazan fumarate tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 750mg/ time, 4 times/day, oral)
  Interventions: Drug: vonoprazan fumarate + amoxicillin（H-14d)

INTERVENTIONS:
Drug: vonoprazan fumarate + high dose amoxicillin（H-10d） — vonoprazan fumarate 20 mg/time, 2 times/day, oral Amoxicillin 750mg/ time, 4 times/day, oral, for 10d
  Arms: H-VA-dual-10
Drug: vonoprazan fumarate + low dose amoxicillin（L-10d) — vonoprazan fumarate 20 mg/time, 2 times/day, oral Amoxicillin1000mg/ time, 2 times/day, oral, for 10d
  Arms: L-VA-dual-10
Drug: vonoprazan fumarate + amoxicillin（H-14d) — vonoprazan fumarate 20 mg/time, 2 times/day, oral Amoxicillin 750mg/ time, 4 times/day, oral, for 14d
  Arms: H-VA-dual-14

SUMMARY:
Helicobacter pylori infection is closely related to gastritis, peptic ulcer, mucosa-associated lymphoid tissue lymphoma and gastric cancer. Eradication of HP can significantly improve and reduce HP-related diseases. International and domestic guidelines recommend a 10-14 day quadruple regimen containing bismuth as first-line treatment, achieving an eradication rate of more than 80%. However, some disadvantages of these quadruple regimens, such as severe adverse reactions, high medical costs and low compliance, prevent their application in clinical practice. Studies at home and abroad have shown that high-dose proton pump inhibitors combined with amoxicillin can be used as the first-line treatment for HP eradication, with good efficacy and compliance and low rate of adverse reactions. And because it is a single antibiotic therapy, we do not expect this regimen to increase antibiotic resistance rates for HP. The maintenance of gastric PH > 6 is one of the key factors for HP eradication. The acid inhibition effect of proton pump mainly depends on the degree of individual metabolism of proton pump. Vonoprazan fumarate, a new competitive potassium acid blocker, is not affected by gene polymorphism, and has the advantage of stronger and longer inhibition effect on gastric acid compared with proton pump inhibitors. In most parts of China, HP is characterized by high infection rate and antibiotic resistance rate, requiring higher eradication rate and safety regimen.This study aimed to evaluate two different amoxicillin dosages

(1 g b.i.d. vs. 0.75 g q.i.d.) and two different durations of therapy (14 vs.10 days) to gain insights of the effectiveness of VA dual therapy .

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70, regardless of gender; HP positive in 13C/14C breath test or pathological test; HP eradication has never been performed in the past; Based on the consensus of helicobacter pylori in 2017, it conforms to the HP eradication guideline; The patient voluntarily signed the informed consent.

Exclusion Criteria:

* History of drug allergy in this study; Liver and kidney dysfunction; Cardiopulmonary insufficiency; History of malignant tumor; Taking clopidogrel, warfarin and other drugs simultaneously may affect CYP2C19 metabolism; Pregnant or lactating women; Patients with severe mental illness; Those planning pregnancy; Previous upper gastrointestinal surgery history; Participated in any other clinical investigator in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | 6 week
  Rate of h. pylori successfully eradicated；13C-urea breath testthat will be used to assess this outcome measure

SECONDARY OUTCOMES:
Adverse Event | 6 week
  Rate of adverse event, serious adverse event; Questionnaire that will be used to assess this outcome measure.
Medical financial burden | 6 week
  Medical financial burden；Questionnaire that will be used to assess this outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth afflicated of Sun-yat sen university, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Peng X, Yao JY, Ma YQ, Li GH, Chen HW, Wan Y, Liang DS, Zhang M, Zhi M. Efficacy and Safety of Vonoprazan-Amoxicillin Dual Regimen With Varying Dose and Duration for Helicobacter pylori Eradication: A Multicenter, Prospective, Randomized Study. Clin Gastroenterol Hepatol. 2024 Jun;22(6):1210-1216. doi: 10.1016/j.cgh.2024.01.022. Epub 2024 Feb 1. PMID 38309492